CLINICAL TRIAL: NCT06339502
Title: The Effect of the Use of Jigsaw Technique on Nursing Students' Critical Article Reviews and Students' Opinions on the Technique- Quasi-Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Duzce-U-merve0002
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Education, Distance; Students, Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): With the students in the control group, a standard individual article review will be conducted under the supervision of the instructor.
- Experimental group (Experimental): The students in the experimental group will be divided into 7 main groups of 7 students according to their academic grade point average. In these groups, each member will be responsible for one of the 7 sections of the article. Those who take the same section in the groups will unite to form expert groups and specialize by working on this section. Students will then return to their main groups and analyze an experimental article. From the groups presenting their reviews, a winner will be selected.
  Interventions: Behavioral: Jigsaw Technique

INTERVENTIONS:
Behavioral: Jigsaw Technique — The jigsaw technique is one of the cooperative learning methods. A topic planned to be learned in the lesson is divided into sections and these sections are distributed to the students in the main group. Students who are responsible for the same sections in the groups combine to form expert groups and specialize by working on the subject. They then return to their main group to share their knowledge and make a presentation on the topic.
  Arms: Experimental group

SUMMARY:
Studies have proven that the Jigsaw learning method, one of the innovative learning methods, is an effective educational learning tool for nursing students. For nursing education to be sufficient to provide students with the modern roles required by the profession, students must actively learn instead of a memorized undergraduate education. -Training programs should enable them to participate in the teaching process. One of these programs is cooperative learning methods. The jigsaw learning technique creates a contemporary learning model by creating a positive learning environment, individualizing students and developing a sense of responsibility. No scientific literature has been found regarding the effect of the Jigsaw learning method on teaching critical article reading skills in nursing research courses in nursing education. It is assumed that the data obtained in this study will contribute to the effect of critical article reading training given using the Jigsaw technique, one of the cooperative learning techniques in nursing education, on students' critical article reviews and opinions about the technique.

DETAILED DESCRIPTION:
Studies have proven that the Jigsaw learning method, one of the innovative learning methods, is an effective educational learning tool for nursing students. For nursing education to be sufficient to provide students with the modern roles required by the profession, students must actively learn instead of a memorized undergraduate education. -Training programs should enable them to participate in the teaching process. One of these programs is cooperative learning methods. The jigsaw learning technique creates a contemporary learning model by creating a positive learning environment, individualizing students and developing a sense of responsibility. No scientific literature has been found regarding the effect of the Jigsaw learning method on teaching critical article reading skills in nursing research courses in nursing education. It is assumed that the data obtained in this study will contribute to the effect of critical article reading training given using the Jigsaw technique, one of the cooperative learning techniques in nursing education, on students' critical article reviews and opinions about the technique.

Aim: The purpose of the study is to determine the effect of using the Jigsaw technique on nursing students' critical article reviews and the student's opinions about the technique.

Method: This is a randomized-controlled experimental study. The study will be carried out in the Spring Semester of the 2023-2024 Academic Year, with the students who attend the Research in Nursing Course at the Nursing Department of the Faculty of Health Sciences of Düzce University. The universe is the students taking the Research in Nursing course (191 people). To obtain a statistically significant difference with a 5% significance level, 80% power, and an effect size of 0.50, a total of 144 individuals will be randomly selected, with the number of people in the experimental and control groups being 2:1. A coin toss will be used to determine the experimental and control groups, and students will be randomly assigned to the groups.

Data accumulation methods: In the study, descriptive features form, critical thinking disposition scale, Kolb's Learning Style Inventory, Self Directed Learning Skills Scales and Jigsaw Opinion Scale will be used as data

Pre-tests will be administered to the students in the control group and individual homework will be given to the students. They will be provided to analyze articles under the supervision of the researcher. Post-tests will be applied.

Students in the experimental group will be administered a pre-test. Students will be heterogeneously divided into eight groups according to their academic grade point average. The groups will consist of 7 people. Each student will be responsible for one of the 7 article sections. These sections are: 1) Title

- Abstract 2) Introduction 3) Method 4) Results 5) Discussion 6) Conclusion and Recommendations 7) Limitations - Resources. Within the group, it will be determined which member will be responsible for which article section. collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Students must volunteer to participate in the study.

Exclusion Criteria:

* Students who decline to participate in the study
* Students who will not be able to participate in the application continuously

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
Critical Thinking Disposition Scale | 28 to 30 days
  Critical Thinking Disposition Scale: The scale was developed by Semerci in 2000. The scale consists of 49 items with 5 dimensions. Sub-themes of the scale are metacognition, flexibility, systematicity, tenacity-patience and open-mindedness. 14 of the items are in metacognition, 11 of these are in flexibility, 11 of these are in tenacity and patience, and 8 of these are in open-mindedness. The Cronbach Alpha coefficient of the CDTH is 0.96.
The Kolb Learning Style Inventory-III | 28 to 30 days
  Although the expression changes were made to concretize the inventory, the last version of which was prepared in 1999, the important difference is in the evaluation and coding processes.In addition, in the final version of the scale, the style names were changed to "Decomposition", "Switching", "Assimilation" and "Accommodation". Kolb describes this change as "a small but important change".This difference comes to the fore during the interpretation of the scale. The scale includes 12 complementary items, as in the previous version. The four options in each item are scored between 1 and 4. The lowest score from the scale is 12, the highest score is 48.
Self Directed Learning Skills Scale | 28 to 30 days
  The scale was developed by Tekkol and Demirel (2018). "Self-Directed Learning Skills Scale" consists of 21 items and four dimensions. Dimensions of the scale; named as motivation, self-monitoring, self-control and self-confidence.The Cronbach Alpha internal consistency coefficient was 0,895.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Cakar, PhD, Principal Investigator — Duzce University
Locations (2):
- Turkey (Türkiye) (2):
  - Duzce University, Düzce
  - Düzce University, Düzce